CLINICAL TRIAL: NCT00608062
Title: Biological Mechanisms of Arterial Stiffening With Age and Estrogen Deficiency
Brief Title: Sex Hormones and Atherosclerosis Prevention in Perimenopausal Women
Acronym: SHAPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 06-0537; R01AG027678 (NIH)
Record Dates: First submitted 2008-01-31; First posted 2008-02-06 (Estimated); Results first posted 2020-12-24 (Actual); Last update posted 2020-12-24 (Actual); Status verified 2020-12

CONDITIONS: Arterial Stiffening; Aging; Menopause
Keywords: endothelial function; women; female; estrogen deficiency; sex hormones; adiposity; oxidative stress; antioxidants
MeSH Terms: conditions — Obesity | interventions — ganirelix

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Pre1 (Experimental): Premenopausal - GnRHant plus estradiol
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal estradiol patch
- Pre2 (Placebo Comparator): Premenopausal - GnRHant plus placebo
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal placebo patch
- Peri1 (Experimental): Perimenopausal (early) - GnRHant plus estradiol
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal estradiol patch
- Peri2 (Placebo Comparator): Perimenopausal (early) - GnRHant plus placebo
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal placebo patch
- Peri3 (Experimental): Perimenopausal (late) - GnRHant plus estradiol
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal estradiol patch
- Peri4 (Placebo Comparator): Perimenopausal (late) - GnRHant plus placebo
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal placebo patch
- Post1 (Experimental): Postmenopausal - GnRHant plus estradiol
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal estradiol patch
- Post2 (Placebo Comparator): Postmenopausal - GnRHant plus placebo
  Interventions: Drug: GnRHant - Ganirelix acetate; Drug: Transdermal placebo patch

INTERVENTIONS:
Drug: GnRHant - Ganirelix acetate — 1 subcutaneous injection at 0.5 mg then daily injections of 0.25 mg for 6 days (total of 7 days of injections); testing will occur on injection day 4 and day 7
  Other Names: Ganirelix
Drug: Transdermal estradiol patch — 0.075mg/d starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
  Arms: Peri1; Peri3; Post1; Pre1
Drug: Transdermal placebo patch — Starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
  Arms: Peri2; Peri4; Post2; Pre2

SUMMARY:
The purpose of this study is to find out why women's arteries stiffen as they go through menopause, and how this is affected by estrogen loss. We believe that arteries stiffen with the loss of estrogen because of "oxidative stress," the production of molecules that can damage cells and tissues in the body, and because the arteries lose their ability to expand, or dilate.

DETAILED DESCRIPTION:
As women get older and go through menopause, estradiol levels decrease. Also with aging, the arteries that are located around the heart get stiffer. Over time this increase in arterial stiffness can lead to a number of health problems such as high blood pressure and heart disease. In this study we want to find out if a short-term drop in estrogen levels in premenopausal and perimenopausal women can cause arteries to become stiffer, and why this happens. Additionally, in postmenopausal women, we want to find out if a short-term increase in estrogen levels causes their arteries to become more flexible (less stiff).

Arterial health (i.e., stiffness) will be examined in premenopausal, perimenopausal and postmenopausal women before and after they are given a drug called Ganirelix™ (for 7 days), which will markedly lower their reproductive hormones. After the first 4 days of taking Ganirelix™, the women will be randomly placed into 1 of 2 treatment groups to take either estrogen (0.075 mg/d skin patch) replacement or placebo for the rest of the Ganirelix treatment. This is to increase estrogen levels back to the normal level. After having the patch on for 4 days, arterial health will be examined again.

Pre-specified Outcome Measures were divided into unit-of-measurement specific Outcome Measure tables for the purposes of results reporting to ClinicalTrials.gov

ELIGIBILITY:
Inclusion Criteria:

* Healthy women of all races and ethnic backgrounds in one of the following groups:

  * Premenopausal: 18-49 years, regular menstrual cycles with no change in observed cycle length (21-35 days)
  * Perimenopausal: 40-55 years, categorized as either early (at least 2 cycles with cycle length changes of at least 7 days) or late (more than 3 months of amenorrhea) transition
  * Postmenopausal: 45-70 years, more than 12 months of amenorrhea as defined by the menopausal staging system (STRAW); additionally, postmenopausal women will be categorized into early and late stages as defined by the STRAW definition, specifically, women who are less than 5 years postmenopause will be considered early, and women more than 6 years will be categorized as late
* All postmenopausal women will have undergone natural menopause
* No oral contraceptive or Hormone Replacement Therapy (HRT) use for at least 6 months
* Resting blood pressure less than 140/90 mmHg
* Plasma glucose concentrations less than 110 mg/dl under fasting conditions
* Sedentary or recreationally active (less than 3 days of vigorous aerobic exercise)
* No use of medications that might influence cardiovascular function
* Nonsmokers
* No use of vitamin supplements or willing to stop use for duration of the study

Exclusion Criteria:

* History of or active estrogen-dependent neoplasms, acute liver or gallbladder disease, vaginal bleeding, venous thromboembolism, hypertriglyceridemia, and cardiovascular disease
* Known allergy to transdermal patch or GnRHant
* Other contraindications to HRT and GnRHant

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2007-03; Primary Completion 2012-10-25 (Actual); Study Completion 2012-10-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie L Moreau, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Center, Clinical Translational Research Center and Exercise Research Laboratory, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moreau KL, Donato AJ, Seals DR, DeSouza CA, Tanaka H. Regular exercise, hormone replacement therapy and the age-related decline in carotid arterial compliance in healthy women. Cardiovasc Res. 2003 Mar;57(3):861-8. doi: 10.1016/s0008-6363(02)00777-0. PMID 12618248
- [Background] Moreau KL, Gavin KM, Plum AE, Seals DR. Ascorbic acid selectively improves large elastic artery compliance in postmenopausal women. Hypertension. 2005 Jun;45(6):1107-12. doi: 10.1161/01.HYP.0000165678.63373.8c. Epub 2005 May 2. PMID 15867135
- [Background] Virdis A, Ghiadoni L, Pinto S, Lombardo M, Petraglia F, Gennazzani A, Buralli S, Taddei S, Salvetti A. Mechanisms responsible for endothelial dysfunction associated with acute estrogen deprivation in normotensive women. Circulation. 2000 May 16;101(19):2258-63. doi: 10.1161/01.cir.101.19.2258. PMID 10811592
- [Background] Ihionkhan CE, Chambliss KL, Gibson LL, Hahner LD, Mendelsohn ME, Shaul PW. Estrogen causes dynamic alterations in endothelial estrogen receptor expression. Circ Res. 2002 Nov 1;91(9):814-20. doi: 10.1161/01.res.0000038304.62046.4c. PMID 12411396
- [Background] Eskurza I, Monahan KD, Robinson JA, Seals DR. Effect of acute and chronic ascorbic acid on flow-mediated dilatation with sedentary and physically active human ageing. J Physiol. 2004 Apr 1;556(Pt 1):315-24. doi: 10.1113/jphysiol.2003.057042. Epub 2004 Jan 30. PMID 14754992
- [Background] Gavin KM, Jankowski C, Kohrt WM, Stauffer BL, Seals DR, Moreau KL. Hysterectomy is associated with large artery stiffening in estrogen-deficient postmenopausal women. Menopause. 2012 Sep;19(9):1000-7. doi: 10.1097/gme.0b013e31825040f9. PMID 22692329
- [Background] Moreau KL, Meditz A, Deane KD, Kohrt WM. Tetrahydrobiopterin improves endothelial function and decreases arterial stiffness in estrogen-deficient postmenopausal women. Am J Physiol Heart Circ Physiol. 2012 Mar 1;302(5):H1211-8. doi: 10.1152/ajpheart.01065.2011. Epub 2012 Jan 13. PMID 22245769
- [Result] Moreau KL, Hildreth KL, Meditz AL, Deane KD, Kohrt WM. Endothelial function is impaired across the stages of the menopause transition in healthy women. J Clin Endocrinol Metab. 2012 Dec;97(12):4692-700. doi: 10.1210/jc.2012-2244. Epub 2012 Sep 11. PMID 22969140

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from the Denver metro area between March 2007 and March 2012. The first participant was enrolled on March 6, 2007 and the last participant was enrolled in March 2012.
Pre-assignment Details: A total of 155 women consented to participate. During screening, 33 women did not qualify (12 premenopausal, 14 perimenopausal [11 early- and 3 late], and 7 postmenopausal). Twenty-three withdrew from participation before baseline testing and 7 women withdrew from participation after baseline testing but prior to randomization.
Groups:
- Peri1: Perimenopausal (early and late combined) - GnRHant plus estradiol
  GnRHant - Ganirelix acetate: 1 subcutaneous injection at 0.5 mg then daily injections of 0.25 mg for 6 days (total of 7 days of injections); testing will occur on injection day 4 and day 7
  Transdermal estradiol patch: 0.075mg/d starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
- Peri2: Perimenopausal (early and late combined) - GnRHant plus placebo
  GnRHant - Ganirelix acetate: 1 subcutaneous injection at 0.5 mg then daily injections of 0.25 mg for 6 days (total of 7 days of injections); testing will occur on injection day 4 and day 7
  Transdermal placebo patch: Starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
Period: Overall Study
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Started (Randomization to group assignment occurred following GnRHant alone.) | 12 (25 women completed baseline testing, 4 women withdrew prior to randomization) | 12 | 19 (43 women completed baseline testing, 3 women withdrew prior to randomization) | 21 | 13 | 15
Completed | 12 | 12 | 19 | 21 | 13 | 15
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For primary outcome brachial artery FMD, 91 completed the study. Four participants did not have usable FMD data due to poor ultrasound image quality or technical issues with image acquisition; baseline analysis and results for the remaining 87 women are presented.
Groups:
- Peri1: Perimenopausal - GnRHant plus estradiol
  GnRHant - Ganirelix acetate: 1 subcutaneous injection at 0.5 mg then daily injections of 0.25 mg for 6 days (total of 7 days of injections); testing will occur on injection day 4 and day 7
  Transdermal estradiol patch: 0.075mg/d starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
- Peri2: Perimenopausal - GnRHant plus placebo
  GnRHant - Ganirelix acetate: 1 subcutaneous injection at 0.5 mg then daily injections of 0.25 mg for 6 days (total of 7 days of injections); testing will occur on injection day 4 and day 7
  Transdermal placebo patch: Starting on day 4 of the injections following testing time point two; continue for 3 days and retest (day 7)
- Total: Total of all reporting groups
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2 | Total
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13 | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 17 | 21 | 12 | 11 | 85
  >=65 years | 0 | 0 | 0 | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (8) | 33 (7) | 49 (3) | 50 (4) | 56 (5) | 60 (6) | 47 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 17 | 21 | 12 | 13 | 87
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 17 | 21 | 12 | 13 | 87
Body Mass [Mean (Standard Deviation); unit: kg] | 66.8 (15.6) | 64.2 (11.0) | 65.6 (8.1) | 68.7 (11.9) | 70.5 (14.7) | 69.7 (9.3) | 67.6 (11.7)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 23.8 (5.6) | 24.4 (5.3) | 24.1 (3.2) | 25.2 (3.9) | 26.7 (5.9) | 26.5 (2.7) | 25.1 (4.4)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 109 (8) | 110 (7) | 113 (14) | 115 (11) | 117 (14) | 120 (14) | 114 (12)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 70 (7) | 72 (5) | 71 (9) | 73 (6) | 73 (8) | 74 (10) | 72 (8)
VO2peak [Mean (Standard Deviation); unit: ml/kg/min] | 35.3 (6.0) | 31.0 (5.5) | 27.7 (4.0) | 27.5 (5.8) | 24.8 (3.9) | 24.1 (2.9) | 28.2 (5.9)
Glucose [Mean (Standard Deviation); unit: mmol/L] | 4.7 (0.3) | 4.6 (0.6) | 4.5 (0.3) | 4.7 (0.5) | 5.0 (0.7) | 4.6 (0.6) | 4.7 (0.5)
Insulin [Median (Inter-Quartile Range); unit: pmol/L] | 38 [21 to 66] | 42 [30 to 85] | 28 [21 to 66] | 28 [21 to 66] | 28 [21 to 45] | 31 [23 to 82] | 35 [28 to 76]
Total Cholesterol [Mean (Standard Deviation); unit: mmol/L] | 3.7 (0.7) | 4.0 (0.9) | 4.5 (0.9) | 4.2 (0.6) | 4.7 (0.9) | 4.7 (0.9) | 4.3 (0.9)
Low-density Lipoprotein [Mean (Standard Deviation); unit: mmol/L] | 2.3 (0.5) | 2.2 (0.7) | 2.7 (1.0) | 2.4 (0.5) | 2.9 (0.8) | 2.8 (0.9) | 2.6 (0.8)
High-density Lipoprotein [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.1) | 1.3 (0.2) | 1.3 (0.2) | 1.3 (0.3) | 1.3 (0.3) | 1.3 (0.3) | 1.3 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Arterial Stiffness (Carotid Artery Compliance) During Saline
Description: Carotid artery compliance measured by carotid artery ultrasound and brachial artery blood pressure
Time Frame: Baseline, day 4 of GnRHant and day 7 of GnRHant and estradiol or placebo treatment
Population: Early and late perimenopausal were collapsed into 1 perimenopausal group
Measure: Mean (Standard Deviation); unit: mm2/mm Hg×10-1
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 19 | 21 | 13 | 15
mm2/mm Hg×10-1
  Baseline | 1.31 (0.27) | 1.34 (0.18) | 0.90 (0.27) | 1.02 (0.33) | 0.89 (0.25) | 0.74 (0.23)
  GnRHant alone: number analyzed (Participants) | 11 | 11 | 19 | 20 | 13 | 15
  GnRHant alone | 1.27 (0.27) | 1.19 (0.34) | 0.89 (0.27) | 0.94 (0.29) | 0.85 (0.24) | 0.79 (0.22)
  GnRHant + Add-Back | 1.29 (0.26) | 1.14 (0.38) | 0.98 (0.27) | 0.94 (0.27) | 0.92 (0.27) | 0.80 (0.19)

2. Primary Outcome: Endothelial Function
Description: Brachial artery flow-mediated dilation (FMD) assessed by ultrasound. This other outcome measure was originally specified as "Secondary" in error and has been updated to "Primary" to be consistent with the protocol.
Time Frame: Baseline, day 4 of GnRHant and Day 7 of GnRHant and estradiol or placebo treatment
Population: Numbers for some groups are reduced because of poor ultrasound image quality.
Measure: Mean (Standard Deviation); unit: % Diameter Change
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
% Diameter Change
  Baseline | 9.8 (2.5) | 11.3 (2.5) | 7.7 (2.6) | 6.1 (2.7) | 5.4 (1.7) | 5.3 (2.2)
  Day 4 of GnRHant alone | 7.1 (2.3) | 8.9 (2.7) | 5.8 (2) | 6.6 (2) | 4.9 (1.5) | 4.9 (1.4)
  Day 7 of GnRHant plus treatment: number analyzed (Participants) | 11 | 12 | 17 | 21 | 11 | 11
  Day 7 of GnRHant plus treatment | 10.6 (3.3) | 7.8 (3.0) | 9.6 (3.3) | 6.1 (2.7) | 8.4 (2.4) | 4.2 (1.7)
  Acute Vitamin C Infusion Day 7: number analyzed (Participants) | 12 | 9 | 17 | 20 | 9 | 9
  Acute Vitamin C Infusion Day 7 | 8.4 (3.1) | 11.2 (4.8) | 9.3 (3.4) | 11.2 (3.6) | 7.8 (3.4) | 6.7 (2.8)
Statistical Analysis 1: Comparison: Pre1 vs Pre2 vs Peri1 vs Peri2 vs Post1 vs Post2; Test type: Other — Repeated measurements of FMD were modeled using a general linear mixed model with maximum likelihood estimation. An unstructured covariance structure allowing for heterogeneity in the parameter estimate for each level of menopause stage was chosen for the model based on using AIC to compare various covariance structures; p = 0.05, Mixed Models Analysis

3. Other Pre Specified Outcome: Supine Brachial Blood Pressures
Time Frame: Baseline, day 4 of GnRHant and day 7 of GnRHant and estradiol or placebo treatment
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
mmHg
  Baseline | 102 (10) | 108 (9) | 111 (13) | 109 (15) | 117 (10) | 123 (13)
  Day 4 of GnRHant alone | 107 (7) | 111 (13) | 112 (12) | 108 (13) | 116 (9) | 115 (8)
  Day 7 of GnRHant plus treatment | 103 (10) | 110 (14) | 108 (13) | 109 (16) | 112 (10) | 111 (8)

4. Other Pre Specified Outcome: Estradiol
Description: This other outcome measure was originally specified as "Secondary" in error and has been updated to "Other, Pre-specified" to be consistent with the protocol. Serum estradiol for clinical characteristics and to detect changes in estradiol levels with the interventions.
Time Frame: Baseline, day 4 of GnRHant and day 7 of GnRHant and estradiol or placebo treatment
Population: Data are for subsample of women who completed FMD with useuable data
Measure: Median (Inter-Quartile Range); unit: pmol/L
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
pmol/L
  Baseline | 229 [117 to 332] | 270 [128 to 484] | 360 [46 to 508] | 147 [62 to 316] | 39 [37 to 49] | 37 [37 to 42]
  GnRHant alone | 147 [87 to 183] | 127 [96 to 243] | 92 [37 to 468] | 99 [37 to 321] | 37 [37 to 42] | 37 [37 to 42]
  GnRhant+Add-back | 202 [140 to 481] | 134 [117 to 183] | 187 [81 to 569] | 106 [37 to 321] | 165 [128 to 223] | 37 [37 to 39]
Statistical Analysis 1: Comparison: Pre1 vs Pre2 vs Peri1 vs Peri2 vs Post1 vs Post2; Test type: Other — Similar analyses as primary outcome; p = 0.05, Mixed Models Analysis

5. Other Pre Specified Outcome: Progesterone
Description: This other outcome measure was originally specified as "Secondary" in error and has been updated to "Other, Pre-specified" to be consistent with the protocol. Serum progesterone was measured for clinical characteristics and to determine changes in sex hormones.
Time Frame: Baseline, Day 4 GnRHant, Day 7 GnRHant+Add-back
Population: Data presented are from those women who had FMD with usable images
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
nmol/L
  Baseline | 1.8 [0.7 to 2.5] | 2.1 [1.0 to 3.1] | 1.1 [0.6 to 1.9] | 1.3 [1.0 to 1.9] | 1.1 [0.6 to 1.3] | 0.9 [0.6 to 1.3]
  GnRHant alone | 1.3 [0.4 to 2.9] | 1.7 [0.7 to 3.7] | 1.0 [0.6 to 1.9] | 1.0 [0.6 to 2.5] | 1.0 [0.3 to 1.3] | 0.6 [0.3 to 1.1]
  GnRhant+Add-back | 1.0 [0.5 to 2.7] | 1.0 [0.6 to 2.1] | 0.8 [0.6 to 3.6] | 1.6 [0.7 to 4.9] | 1.0 [0.6 to 1.0] | 0.6 [0.6 to 1.1]
Statistical Analysis 1: Comparison: Pre1 vs Pre2 vs Peri1 vs Peri2 vs Post1 vs Post2; Test type: Other — same analysis as primary outcome; p = 0.05, Mixed Models Analysis

6. Other Pre Specified Outcome: Total Antioxidant Status (TAS)
Description: This other outcome measure was originally specified as "Secondary" in error and has been updated to "Other, Pre-specified" to be consistent with the protocol. TAS is an antioxidant and is a biomarker of oxidative stress.
Time Frame: Baseline, Day 4 GnRHant, Day 7 GnRHant+Add-back
Population: Data are presented from participants that completed the endothelial function testing and who had usable images.
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
nmol/L
  Baseline | 1.4 (0.2) | 1.4 (0.2) | 1.3 (0.2) | 1.3 (0.1) | 1.3 (0.2) | 1.3 (0.2)
  GnRHant alone | 1.4 (0.2) | 1.5 (0.1) | 1.3 (0.2) | 1.3 (0.2) | 1.3 (0.1) | 1.4 (0.3)
  GnRhant+Add-back | 1.4 (0.1) | 1.4 (0.1) | 1.3 (0.1) | 1.3 (0.1) | 1.3 (0.2) | 1.3 (0.2)

7. Other Pre Specified Outcome: Endothelin-1 (ET-1)
Description: This other outcome measure was originally specified as "Secondary" in error and has been updated to "Other, Pre-specified" to be consistent with the protocol.
Time Frame: Baseline, Day 4 GnRHant, Day 7 GnRHant+Add-back
Population: Data are presented from women who completed endothelial function testing and whom had usable images
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
pg/mL
  Baseline | 5.2 (1.5) | 5.2 (0.9) | 5.9 (1.3) | 6.2 (1.6) | 6.2 (1.4) | 6.4 (1.1)
  GnRHant alone | 5.5 (1.7) | 5.5 (0.9) | 6.0 (1.8) | 5.9 (0.9) | 6.5 (2.1) | 6.5 (0.9)
  GnRhant+Add-back | 6.0 (1.1) | 5.0 (0.7) | 5.9 (1.6) | 5.7 (1.9) | 6.0 (1.8) | 6.4 (0.9)

8. Other Pre Specified Outcome: Plasma Norepinephrine
Description: as for outcome 7
Time Frame: Baseline, Day 4 GnRHant, Day 7 GnRHant+Add-back
Population: Data are presented from women who completed endothelial function testing and whom had useable images.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
Number analyzed (Participants) | 12 | 12 | 17 | 21 | 12 | 13
pg/mL
  Baseline | 161 [108 to 230] | 184 [101 to 217] | 227 [168 to 280] | 247 [164 to 295] | 231 [127 to 349] | 242 [228 to 331]
  GnRHant alone | 144 [116 to 164] | 156 [103 to 252] | 235 [183 to 282] | 233 [159 to 341] | 280 [156 to 362] | 217 [180 to 282]
  GnRhant+Add-back | 146 [118 to 214] | 217 [152 to 282] | 231 [168 to 295] | 217 [152 to 282] | 204 [168 to 280] | 221 [162 to 303]

ADVERSE EVENTS:
Description: Participants were asked at each vascular visit to complete a symptom questionnaire. These data were reviewed immediately by the PI and the study physician. Further, these data were summarized for the Safety Officer annually.
Arm/Group | Pre1 | Pre2 | Peri1 | Peri2 | Post1 | Post2
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/19 | 0/21 | 0/13 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/19 | 0/21 | 0/13 | 0/15
Other Adverse Events (participants affected / at risk) | 8/12 | 4/12 | 9/19 | 8/21 | 5/13 | 4/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pre1 (N=12) | Pre2 (N=12) | Peri1 (N=19) | Peri2 (N=21) | Post1 (N=13) | Post2 (N=15)
Cardiovascular/neurology (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) — Vasal vagal to nitrogylcerine
Bloating (Gastrointestinal disorders) | 2 (2) | 1 (1) | 4 (4) | 2 (2) | 2 (2) | 1 (1)
Breast tenderness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Injection site reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 2 (2) — Dermatology
Joint Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Patch irritation (Skin and subcutaneous tissue disorders) | 6 (6) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 2 (2) — Transdermal patch irritation, redness
Vaginal bleeding (Reproductive system and breast disorders) | 4 (4) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Other urogenital (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1) — Vaginal discharge, dryness

LIMITATIONS AND CAVEATS:
Budget cuts lead to: 1) endothelial cell protein expression outcome not analyzed and deleted; 2) small numbers of early and late perimenopausal groups, thus, it was collapsed into 1 peri group. Ultrasound image quality also lead to small numbers.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No